CLINICAL TRIAL: NCT04889794
Title: GPS Project - Evaluation of the Impact of the Reorganization of Work Into a Family Medicine Group on Pharmacotherapy and Support for the Autonomy of Seniors With Major Neurocognitive Disorders
Brief Title: GPS Project Evaluation of the Impact of the Reorganization of Work Into a Family Medicine Group on Pharmacotherapy and Support for the Autonomy of Seniors With Major Neurocognitive Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: CISSS de Chaudière-Appalaches (Other Government); Ciusss de L'Est de l'Île de Montréal (Other); Fonds de la Recherche en Santé du Québec (Other Government)
Responsible Party: Principal Investigator, Dre Edeltraut Kröger, Professor, CHU de Quebec-Universite Laval
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MP-23-2020-732 - GPS
Record Dates: First submitted 2021-05-12; First posted 2021-05-17 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Major Neurocognitive Disorder
Keywords: living lab; major neurocognitive disorder; polypharmacy; health outcomes; pharmacists; home care; family medicine groups; deprescribing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposed FMGs to GPS intervention (Experimental): Patients who are followed by FMGs exposed to the GPS intervention. They will receive the GPS intervention.
  Interventions: Other: GPS clinical intervention
- Non exposed FMGs to GPS intervention (No Intervention): Patients who are part of the FMGs not exposed to the GPS intervention. They will receive the usual care and services.

INTERVENTIONS:
Other: GPS clinical intervention — Nurses and doctors in exposed FMGs and home care teams (HCTs) will be asked to refer to the FMG pharmacist all seniors undergoing cognitive evaluation OR referred to a memory clinic OR recently diagnosed with a cognitive disorder, for a complete and critical review of their medication therapy. FMG pharmacists will be asked to conduct an interview with each referred senior and his or her caregiver, if applicable, in order to establish the best possible treatment regimen. They will compare the information collected with another reliable data source (e.g., pharmacy records) in order to perform medication reconciliation and will then evaluate the medication related problems. Pharmacist will establish a care plan and the follow-ups to be carried out with the patient in collaboration with the health care team. There will be no drug or devices tested, it is a human clinical intervention by a pharmacist.
  Arms: Exposed FMGs to GPS intervention

SUMMARY:
The model of care tested in the GPS project aims to optimize pharmacotherapy for seniors undergoing cognitive assessment or suffering from major neurocognitive disorder (MCND) at home. The goal is to reduce polymedication, inappropriate medications and the treatment burden of seniors and to maintain their cognitive health, quality of life and autonomy. The intervention will include knowledge exchange sessions with nurses, pharmacists, and doctors in FMGs, and increased collaboration between these professionals and home care services teams. Other goal is to increase the satisfaction of the seniors, their families, and the professionals involved in the GPS project.

DETAILED DESCRIPTION:
: The GPS project is part of the desire to keep seniors with major neurocognitive disorder (MCND) in their homes for as long as possible. Medication can contribute to cognitive loss in seniors and affect their functional autonomy. The arrival of pharmacists in FMGs and the expansion of their practice is opening up new opportunities to promote interdisciplinary collaboration and optimize pharmacotherapy for seniors. During the project, a new model of care, called GPS, is being tested with seniors. A group of seniors (approximately 200) will receive the new care team's new interventions in the FMGs in the "intervention" group. Another group of seniors (about 200) will receive the usual care in other FMGs that will serve as a "control" group. By comparing the results of the two groups, it will be possible to evaluate the effects of new interventions. A period of 12 months will be allocated for the inclusion of seniors. The follow-up of each senior will be approximately 6 months.

ELIGIBILITY:
Inclusion Criteria:

* All seniors (65 years of age or older) undergoing cognitive evaluation OR referred to a memory clinic OR having been diagnosed with cognitive impairment within the last year OR with MCND and followed up at home AND,
* referred to the pharmacist, for the FMGs exposed
* taking prescription medications

Exclusion Criteria:

* Seniors in palliative care OR
* unable to answer questionnaires in French AND without a caregiver.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-09-27 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in number of prescribed medications | Baseline, 3 months and 6 months after inclusion in the study.
  The total number of prescribed medications and 2) the number of potentially inappropriate medications (PIMs) according to the Beers criteria or according to the OptimaMed criteria for participants with advanced MCND will be measured in both groups, before, during and after the study.

SECONDARY OUTCOMES:
Change in treatment burden | Baseline and 6 months follow-up
  The treatment burden level will be measured with the 13-item Multimorbidity Treatment burden questionnaire in the intervention and control groups before and after the study. Each item will be scored as follows: zero (not difficult/ does not apply), one (a little difficult), two (quite difficult), three (very difficult), four (extremely difficult).Scores will be interpreted as suggested by the authors of the original MTBQ instrument: no burden (score 0), low burden (score <10), medium burden (10-22), high burden (>=22)

OTHER OUTCOMES:
Change in number of hospitalizations | 12 months prior to the start of the intervention and in the 12 months afterwards
  The number of hospitalizations in the 12 months prior to the start of the intervention and in the 12 months afterwards will be evaluated by the exploration of the RAMQ data record with the consent of the participant in the intervention and control groups
Change in number of emergency room visits | 12 months prior to the start of the intervention and in the 12 months afterwards
  The number of emergency room visits in the 12 months prior to the start of the intervention and in the 12 months afterwards will be evaluated by the exploration of the RAMQ data record with the consent of the participant in the intervention and control groups.
Change in quality of life | Baseline and 6 months follow-up
  The measure of quality of live will be perform two times with the EQ-5D-5L in the intervention and control groups before and after the study. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. Responses are coded as single-digit numbers expressing the severity level selected in each dimension. For instance, 'slight problems' is always coded as '2'. The digits for the five dimensions can be combined in a 5-digit code that describes the respondent's health state. For example, 21111 means slight problems in the mobility dimension and no problems in any of the other dimensions.

CONTACTS AND LOCATIONS:
Overall Officials: Line Guénette, Ph.D, Study Director — CHU de Québec-Université Laval, Laval University
Locations (2):
- Canada (2):
  - GMF Bordeaux-Cartierville, Montreal, Quebec
  - GMF Abénakis, Saint-Georges, Quebec

REFERENCES:
- [Derived] Guenette L, Kroger E, Bonnan D, Maheu A, Morin M, Belanger L, Vedel I, Wilchesky M, Sirois C, Durand E, Couturier Y, Sourial N, Dallaire C. Reorganizing Pharmaceutical Care in Family Medicine Groups for Older Adults With or at Risk of Major Neurocognitive Disorders: Protocol for a Mixed Methods Study. JMIR Res Protoc. 2022 Nov 17;11(11):e42577. doi: 10.2196/42577. PMID 36264995